CLINICAL TRIAL: NCT01405469
Title: Endoscopic Peroral Myotomy for Treatment of Achalasia: Pilot Study
Brief Title: Endoscopic Peroral Myotomy for Treatment of Achalasia
Acronym: POEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKE Hamburg Endoscopy PV3725
Record Dates: First submitted 2011-05-26; First posted 2011-07-29 (Estimated); Results first posted 2014-12-02 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Achalasia
Keywords: Achalasia; Heller myotomy; Dysphagia; Peroral Endoscopic Myotomy
MeSH Terms: conditions — Esophageal Achalasia; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Peroral Endoscopic Myotomy (Experimental): Patients with achalasia who are designed to either get balloon dilatation or have botulinum toxin injection, or to have surgical intervention (Heller myotomy)for treatment
  Interventions: Other: Peroral Endoscopic Myotomy

INTERVENTIONS:
Other: Peroral Endoscopic Myotomy — A forward-viewing upper endoscope is used with a transparent distal cap attachment. Carbon dioxide gas is necessary for insufflation during the procedures. An endoscopic knife is used to access the submucosa, dissect the submucosal tunnel and also to divide circular muscle bundles over a length of approximately 10cm, extending 2-3cm onto the cardia. An electric generator is used with spray coagulation mode. A coagulating forceps is used for hemostasis as needed. Closure of the mucosal entry site is performed using standard endoscopic clips

SUMMARY:
This study intends to investigate the feasibility, safety and efficacy of peroral endoscopic myotomy for the treatment of achalasia in a single center setting in Europe.

DETAILED DESCRIPTION:
This pilot study intends to investigate the feasibility, safety and efficacy of peroral endoscopic myotomy for the treatment of achalasia in a single center setting in Europe.

16 patients are enrolled to evaluate feasibility, safety and efficacy of peroral endoscopic myotomy. Main outcome measurement is the eckhardt symptom score 3 month after therapy.

Primary outcome:

-eckhardt symptom score 3 month after therapy.

Secondary outcomes:

* Lower esophageal sphincter pressure at 3 month after therapy.
* Reflux symptoms at 3 month after therapy.

For this prospective study, inclusion criteria are achalasia, as diagnosed by established methods (contrast fluoroscopy, manometry, esophagal-gastro-duodenoscopy) and age greater than 18 years. Previous therapy, such as esophageal surgery or previous myotomy are exclusion criterion.

A forward-viewing upper endoscope is used with a transparent distal cap attachment. Carbon dioxide gas is necessary for insufflation during the procedures. An endoscopic knife is used to access the submucosa, dissect the submucosal tunnel and also to divide circular muscle bundles over a length of approximately 10cm, extending 2-3cm onto the cardia. An electric generator is used with spray coagulation mode. A coagulating forceps is used for hemostasis as needed. Closure of the mucosal entry site is performed using standard endoscopic clips.

ELIGIBILITY:
Inclusion criteria:

* Patient with symptomatic achalasia and pre-op barium swallow, manometry and esophagal-gastro-duodenoscopy which are consistent with the diagnosis
* persons of age > 18 years with medical indication for surgical myotomy or Endoscopic balloon dilatation
* Signed written informed consent.

Exclusion criteria:

* Patients with previous surgery of the stomach or esophagus
* Patients with known coagulopathy
* Previous achalasia-treatment with surgery
* Patients with liver cirrhosis and/or esophageal varices
* Active esophagitis
* Eosinophilic esophagitis
* Barrett's esophagus
* Pregnancy
* Stricture of the esophagus
* Malignant or premalignant esophageal lesion
* Candida esophagitis
* Hiatal hernia > 2cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Roesch, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Klinik für Interdisziplinäre Endoskopie, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inoue H, Minami H, Kobayashi Y, Sato Y, Kaga M, Suzuki M, Satodate H, Odaka N, Itoh H, Kudo S. Peroral endoscopic myotomy (POEM) for esophageal achalasia. Endoscopy. 2010 Apr;42(4):265-71. doi: 10.1055/s-0029-1244080. Epub 2010 Mar 30. PMID 20354937
- [Result] von Renteln D, Inoue H, Minami H, Werner YB, Pace A, Kersten JF, Much CC, Schachschal G, Mann O, Keller J, Fuchs KH, Rosch T. Peroral endoscopic myotomy for the treatment of achalasia: a prospective single center study. Am J Gastroenterol. 2012 Mar;107(3):411-7. doi: 10.1038/ajg.2011.388. Epub 2011 Nov 8. PMID 22068665
- See also: University Hospital Hamburg-Eppendorf, Endoscopy Department — http://www.uke.de/kliniken/endoskopie/index.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with symptomatic achalasia
Pre-assignment Details: 16 patients were included as per protocol, no patient was lost during follow-up over a 2 year period
Groups:
- POEM Patients: pilot group of achalasia patients who received POEM Treatment: Endoscopic Myotomy of the Lower Esophageal Sphincter
Period: Overall Study
Arm/Group | POEM Patients
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- POEM Patients: pilot study, first 16 patients who received POEM for treatment of achalasia
Arm/Group | POEM Patients
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (16.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Region of Enrollment [Number; unit: participants]
  Germany | 16

OUTCOME MEASURES:

1. Secondary Outcome: mmHg of the Lower Esophageal Sphincter 3 Months After POEM Procedure
Description: esophageal manometry is done 3 months after POEM procedure to evaluate resting lower esophageal sphincter pressure
Time Frame: manometry at 3 month after therapy
Population: Pilot study group to evaluate feasibility and safety of POEM procedure before initiating studies evaluating long-term efficacy.Patients with primary achalasia, diagnosed by established methods(contrast fluoroscopy, manometry, esophagogastroduodenoscopy(EGD)) and age greater than 18 years were included.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- POEM Patients: pilot group of achalasia patients who received POEM treatment
Arm/Group | POEM Patients
Number analyzed (Participants) | 16
mmHg | 11.8 (9.016200316)

2. Secondary Outcome: Number of Participants With Reflux Symptoms
Description: Number of Participants with Reflux Symptoms during procedure, and 3 and 6 months, and 1, 2 and 5 years after treatment
Time Frame: during procedure, and 3 and 6 months, and 1, 2 and 5 years after treatment
Measure: Number; unit: participants
Arm/Group | POEM Patients
Number analyzed (Participants) | 16
participants | 1

3. Primary Outcome: Treatment Success Defined as Symptom Relief 3 Months After Treatment Based on an Eckhardt Score ≤ 3
Description: eckhardt score is a score to evaluate achalasia discomfort in patients. Patients are being interrogated for dysphagia, regurgitation, and retrosternal pain , correlated with the time frame of occurrence. "with every meal" giving 3 points," daily" (2 points), "sometimes" (1 Point) or "no" (0 Points), as well as weight loss,(>10 kg= 3 points, 5-10 kg=2 points, 0-5 kg=1 point, None=0 points. Scale range is from 0 Points (no achalasia) up to 12 points for the worst achalasia symptoms.
Time Frame: 3 months after treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Eckardt Score
Arm/Group | POEM Patients
Number analyzed (Participants) | 16
Eckardt Score
  symptom relief 3 months after treatment | 1.4 (2.217355783)
  eckhardt score baseline | 8.8 (1.28)
Statistical Analysis 1: Comparison: POEM Patients; this pilot study was created ro evaluate sample size for the following multicenter study, based on manometric outcomes. Mean values between baseline and follow-up were compared using Student ' s t -test for paired samples. P values less then 0.05, two-sided, were considered significant.R 2.13.1(R Development Core Team (2011). Subgroups (partial vs. complete myotomy) were compared using an analysis of variance test adjusted for initial values; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; Mean Difference (Net) = -7.44, Standard Deviation 2.66

4. Secondary Outcome: Number of Participants With Procedure-related Adverse Events
Description: procedure-related adverse events per protocol
Time Frame: procedure to 3 months post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | POEM Patients
Number analyzed (Participants) | 16
Participants | 2

5. Secondary Outcome: Medication 3 Months After POEM
Description: proton pump inhibitor (PPI) use at 3 months after POEM procedure
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | POEM Patients
Number analyzed (Participants) | 16
participants | 1

6. Secondary Outcome: Duration Time Procedure
Description: duration time of POEM procedures in minutes
Time Frame: procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | POEM Patients
Number analyzed (Participants) | 16
minutes | 114 (37.48238475)

7. Secondary Outcome: Days Duration Hospitalization
Description: participants were followed for the duration of hospital stay, an average of 4 days
Time Frame: days of hospitalization for POEM procedure, an average of 4 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | POEM Patients
Number analyzed (Participants) | 16
days | 4.5625 (0.892094913)

8. Secondary Outcome: cm Myotomy Length
Description: myotomy length in cm
Time Frame: POEM procedure
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | POEM Patients
Number analyzed (Participants) | 16
cm | 12 (2.704933764)

9. Secondary Outcome: Percentage of Participants Who Achieved Treatment Success 3 Months After Treatment
Description: eckhardt score is a score to evaluate achalasia discomfort in patients. Patients are being interrogated for dysphagia, regurgitation, and retrosternal pain , correlated with the time frame of occurrence. "with every meal" giving 3 points," daily" (2 points), "sometimes" (1 Point) or "no" (0 Points), as well as weight loss,(>10 kg= 3 points, 5-10 kg=2 points, 0-5 kg=1 point, None=0 points. Scale range is from 0 Points (no achalasia) up to 12 points for the worst achalasia symptoms. Post-myotomy eckhardt score ≤ 3 n individuals has been reached in 15 individuals.
Time Frame: 3 months after treatment
Population: as for outcome 1
Measure: Number; unit: percentage of treated patients
Arm/Group | POEM Patients
Number analyzed (Participants) | 16
percentage of treated patients | 94

ADVERSE EVENTS:
Time Frame: 2 days after POEM
Description: 1 cm superficial ulcer (Forrest III) at the cardia
Arm/Group | POEM Patients
Serious Adverse Events (participants affected / at risk) | 2/16
Other Adverse Events (participants affected / at risk) | 1/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | POEM Patients (N=16)
1 cm superficial ulcer (Forrest III) (Gastrointestinal disorders) | 1 (1) — a 1 cm superficial ulcer (Forrest III) at the cardia was detected on routine EGD, 2 days after POEM.
ulcer in the distal esophagus (Gastrointestinal disorders) | 1 (1) — retrosternal pain 3 weeks after POEM. EGD demonstrated an ulcer in the distal esophagus(FIII). The ulcer was clipped
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | POEM Patients (N=16)
treatment failure (Gastrointestinal disorders) | 1 (1) — eckhardt score 9 three months after POEM

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes